CLINICAL TRIAL: NCT05482217
Title: The Effectiveness of Psychoeducation and Problem-solving (Life-steps) on Depression and Treatment Adherence in HIV Infected Adolescents: an Exploratory Randomized Controlled Trial
Brief Title: The Effectiveness of CBI on Depression and Adherence in HIV Infected Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Botswana (Other)
Collaborators: University of KwaZulu (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UBotswana
Record Dates: First submitted 2022-05-12; First posted 2022-08-01 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-05

CONDITIONS: Medication Nonadherence; Depression; HIV Infections
Keywords: psychoeducation; problem-solving; depression; Life-steps; HIV-infected adolescents; clinical trial
MeSH Terms: conditions — Medication Adherence; Depression; HIV Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): This group was exposed to psychoeducational and problem-solving sessions for five weeks.
  Interventions: Behavioral: Psychoeducation, problem solving and rehearsal (cognitive behavioural intervention)
- The control group (No Intervention): No intervention was given: only the regular clinic advice for five weeks or treatment as usual.

INTERVENTIONS:
Behavioral: Psychoeducation, problem solving and rehearsal (cognitive behavioural intervention) — The highlights of the intervention.
  Session 1: Rapport building and knowledge of HIV
  Session 2: Identifying and Dealing with barriers to good adherence
  Session 3: Identifying and dealing with problems in relation to depression and adherence:
  Session 4: Identifying and dealing with negative cognitions, handling privacy, accessing social Support, and adjusting to HIV and antiretroviral treatment
  Session 5: Rehearsal of practical tips on adherence, handling slips, and strategies to improve quality of life.
  All sessions involved brief periods of relaxation, homework, and a homework review. The last session was concluded with the assessment of satisfaction with the program. The programs were conducted for 60 minutes weekly for five weeks.
  They were delivered by a trained lay counselor and supervised by the principal investigator for five weeks.
  Other Names: Cognitive behavioural intervention (CBI)
  Arms: Intervention group

SUMMARY:
Aim: To explore the effectiveness of psychoeducation and problem-solving (Life-steps) on depression and adherence in HIV-infected adolescents.

Methods: Forty-two adolescents were randomized into 21 controls and 21 intervention groups. The intervention group was exposed to 5-week sessions of life steps applied by a lay counselor. The PHQ-9 and visual analog scale (VAS) were used to measure the outcomes: depression and adherence. They were applied at baseline, 5-weeks, and 24 weeks post-intervention.

DETAILED DESCRIPTION:
General objectives

To explore the effect of psychoeducation and problem solving (LIFE STEPS) technique on medication adherence and depression among mentally ill ALWHIV in Botswana.

Specific Objectives

1. To compare the sociodemographic and clinical variables of the ALWHIV: intervention and control group
2. To explore the effect of psychoeducation and problem solving (LIFE STEPS) on medication adherence and depression among ALWHIV.

Methodology Study Design: Randomised controlled trial to assess the psychological intervention program.

Study sites: The facilities in Gaborone are Baylor children's clinical center of excellence (BCOE), and Princess Marina HIV clinics (PMH).

Subject Population(s) Phase 1: HIV infected adolescents aged, 12 - 19 years.

Subject Recruitment/Sampling Methods:

Using techniques described to determine the sample size for continuous outcome in a randomized controlled trial, a minimum sample size of 25 in each group was calculated to be sufficient to identify a treatment effect of one standard deviation difference in adherence scores based on 5% level of significance and 90% power. A significant treatment effect is expected due to the enormous treatment gap in Africa, such that slight increases by simple interventions will produce huge outcomes. An initial adherence cut-off of less than 95% in VAS visual analog, meeting the criteria for depression on MINI-KID, and a score of 9 and above on PHQ-9 were used for inclusion in the study. Twenty-five participants each were recruited in anticipation of a 25% attrition rate for the intervention and the control groups.

A two-stage random sampling method was adopted to select the participants from the sub-sample of the phase one study. The first stage was to select from those who meet the criteria for the second phase, and the second phase was to allocate the selected sample into two groups randomly. Everyone eligible to participate in the second phase, that is, those who are below the cut-off as earlier alluded to (after the first analysis with SPSS), was given a separate identification number that was linked to their contacts in such a way that their identities (names) were concealed. The sheet that has the identification numbers and contact of the participants was kept separately (locked in a safe cabinet) by the principal investigators (PI). It was only used for follow-up purposes and was destroyed immediately after the study.

The identification numbers of all who are eligible for phase II were entered into the SPSS software, which was used to randomly generate some identification numbers, i.e., 50 participants who were contacted. This process of generating numbers was repeated until 50 participants who are willing to participate were enrolled. These people (with their caregivers) were invited and asked to give their consent/assent after explaining the procedure to them. They were informed about the possibility of being allocated into either an intervention group or control. Those who attended the intervention session and the other group were informed on what to do through their preferred medium of communication. However, the outcome and the detail of the intervention were not discussed with any of the group so as not to introduce a bias. Subsequently, a simple ballot system was used, where folded papers marked with the two choices (intervention = 'I' and control 'C') were presented to all the participants. They were asked to pick one of the folded papers, and the letters they pick indicated which group they belonged to, i.e., 'I' or 'C.' They were informed depending on the letter they pick without telling them the meaning of the letters and the next step to take.

Data Collection Methods Permission was first obtained from the relevant authorities, namely the Ministry of Health and all the health facilities where the recruitment will be done. Written informed consent was obtained from those who have reached the age of consent (18 and 19 years), whereas parental consent and assent were obtained from adolescents below the age of consent (less than 18 years) before commencing the study. This was done by explaining the intention, the benefit, and the risk in an elementary language to all the eligible participants within this age group. Those who refused to agree were exempted from the study regardless of the decisions of their parents or guardians.

A research assistant (RA) was employed and adequately trained in the research instruments and on how to approach the parents and the participants on the clinic days. Specialized training was given on how to obtain information from very young adolescents on sensitive issues. The RA was trained on how to establish rapport, be patient, instill confidence, and be sensitive to their emotional needs. She was trained on how to engage them and when to disengage and or break the interview. A light refreshment was offered within a reasonable limit and without causing an unnecessary inducement.

Fifty adolescents screening positive for depression and poor medication adherence were randomly selected from the first sample (phase I of the study), and randomly allocated into two groups of 25 intervention, and control as alluded to previously. Suitable participants selected from the centers were informed of the objective of the second phase. Their parents were also informed of the plan to psycho-educate them for five weeks. Another consent and or assent were obtained from them before they can be eligible to partake in the second phase.

The participants were made to sit in a small group of five per table, and they were grouped according to their age group into early adolescent (12-14, mid-adolescent (15-17), and late adolescent (18 and above). This enabled the identification of, and attention to the age-specific needs. The meetings were in a comfortable and familiar room that was organized at BCOE. Items such as markers, white paper, paper tape, stickers, a board, a projector, and a computer were supplied. A manualized psychoeducation and problem solving (LIFE STEPS) program on treatment adherence was delivered by a trained lay counselor and supervised by the PI. The program consisted of five structured sessions offered weekly, each lasting 50-60 minutes. The session is basically on identifying problems (such as psychological problems, stigma, and, other related issues), and providing guidance on how to provide adaptive solutions which are age-specific to them.

The sessions were delivered as interactive lectures and small group discussions. They involve interactive discussion, role play, and brief lectures. The plenary sessions which took less than 15 minutes of the sessions were divided majorly into 2 or 3 parts according to the age group, even though they took place concurrently. A few minutes were spent on short relaxation and light exercises. Homework was given after every session. All sessions started with a review of the subject learned in the previous week to allow participants to share how they practiced their skills with the other members of the group. All sessions also started with a brief and simple exercise, such as stretching, clapping, and dancing. At the end of each session, there was also a recapitulation of what had been learned, and new assignments are given to enable participants to practice the new skills. There was a recap of overall sessions based on observations and feedback, where the participants were asked to rate each session on its usefulness and ease of understanding. Transport fares and refreshments were available for the participants.

This rating was on a scale of 1- 10 (1 = not useful or easy to understand, and 10 = very useful or easy to understand also take feedback). Two sessions were randomly selected for audio-recording and were assessed by the supervisor to confirm adherence to the manual. The adherence questionnaires and PHQ-9 were applied at pre-, immediate post-intervention, and 24 weeks. Any change in the level of adherence and depression was measured across groups after exposing the experimental group to five weeks of brief psychological intervention.

Measures Socio-Demographic and Clinical Characteristics Datasheet This subsection consisted of relevant questions on the socio-demographic characteristics of the respondents such as age, religion; ethnicity; position in the family; parent's marital status, educational level, and gender. This also included questions on type and level of social support, clinical variables such as mode of HIV transmission, age at first diagnosis (HIV), previous and current CD4 count, and viral load. Other relevant clinical variables such as frequency of clinic attendance and level of adherence were retrieved from their records with their permission and those of their parents. This section of the questionnaire was designed by the researcher based on a review of previous studies.

MINI-KID MINI-KID is a brief structured clinical diagnostic interview designed to assess the existence of 24 ICD-10 and DSM-IV mental disorders comprehensively and concisely. This interviewer-administered instrument is suitable for adolescents and has been used in various populations, including HIV adolescents in sub-Saharan African settings.

All the instruments were translated into Setswana (the predominant language in Botswana) using the procedure of iterative back-translation by a panel of bilingual experts.

Depression: Patient Health Questionnaire (PHQ-9) is a depression module, which is provisionally used to diagnose depression and grade the severity of symptoms in general medical and mental health settings. It has nine items based on the Diagnostic and Statistical Manual of Mental Disorders, fourth edition (DSM-IV) criteria, and the scores range from "0" (not at all) to "3" (nearly every day). ThePHQ-9 has been validated for use in Botswana. The cutoff of 9 or more is consistent with a diagnosis of a major depressive episode in Botswana and will be used for inclusion in this study.

Data Analysis The study outcomes were depression (measures using PHQ-9) and treatment adherence (VAS). Between groups, comparisons were made based on the intention-to-treat sample. The study collected data for baseline, 5-week, and 24-weeks follow-up. Data from the 24-weeks follow-up was collected from only the intervention group. Wilcoxon rank-sum test was used to assess the differences between the intervention and control groups at various time points when the outcome is in a continuous format. Changes in depression and adherence score over time within assigned groups were assessed using Wilcoxon signed-rank test (if two-time points) and Friedman ANOVA (more than two-time points). The effect size was calculated based on Wilcoxon signed rank where r=|z/√N|. The magnitude was based on Cohen's classification of effect sizes which is 0.1 (small effect), 0.3 (moderate effect), and 0.5 and above (large effect). The relationship between the two outcomes (PHQ-9 and VAS) scores was assessed using Spearman correlation.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected adolescents aged, 12 - 19 years
* On ART for a minimum of six months.
* Speak or communicate in Setswana or English.
* Outpatient
* Willing to participate

Exclusion Criteria:

• Psychotic, and intellectually disabled patients

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2021-07-26 (Actual); Primary Completion 2021-11-02 (Actual); Study Completion 2022-05-03 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms were measured with Patient Health Questionnaire (PHQ-9), has sensitivity and specificity of 0.8 and 0.7. The cut-off of nine or more was consistent with a diagnosis of depression | 5 weeks
  Change in PHQ-9 score or change in depressive symptoms score

SECONDARY OUTCOMES:
Medication adherence: measured with the Visual Analogue Scale (VAS), a horizontal line, 10cm long, and calibrated by 5 from 0 to 100. Score of <95% is suboptimal adherence based on 30 days pill use. It exhibits medium to large strength (r = 0.5-0.7). | 5 weeks
  Change in Visual analogue score or change in medication adherence score

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor children's clinical center of excellence, Gaborone, Botswana

IPD SHARING:
Plan to Share IPD: No
Anonymised data may be shared on request by the publisher

REFERENCES:
- [Derived] Olashore AA, Paruk S, Ogunwale A, Ita M, Tomita A, Chiliza B. The effectiveness of psychoeducation and problem-solving on depression and treatment adherence in adolescents living with HIV in Botswana: an exploratory clinical trial. Child Adolesc Psychiatry Ment Health. 2023 Jan 4;17(1):2. doi: 10.1186/s13034-022-00541-3. PMID 36600262